CLINICAL TRIAL: NCT04595747
Title: Phase 2 Study of Rogaratinib (BAY 1163877) in the Treatment of Patients With Sarcoma Harboring Alterations in Fibroblast Growth Factor Receptor (FGFR) 1-4 and SDH-Deficient Gastrointestinal Stromal Tumor (GIST)
Brief Title: Testing the Anti-cancer Drug, Rogaratinib (BAY 1163877), for Treatment of Advanced Sarcoma With Alteration in Fibroblast Growth Factor Receptor (FGFR 1-4), and in Patients With SDH-deficient Gastrointestinal Stromal Tumor (GIST)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-08011; NCI-2020-08011 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-070; 10411 (Other: Dana-Farber - Harvard Cancer Center LAO); 10411 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2020-10-17; First posted 2020-10-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Gastrointestinal Stromal Tumor; Locally Advanced Sarcoma; Metastatic Gastrointestinal Stromal Tumor; Metastatic Sarcoma; Stage III Gastric and Omental Gastrointestinal Stromal Tumor AJCC v8; Stage III Small Intestinal, Esophageal, Colorectal, Mesenteric, and Peritoneal Gastrointestinal Stromal Tumor AJCC v8; Stage IV Gastric and Omental Gastrointestinal Stromal Tumor AJCC v8; Stage IV Small Intestinal, Esophageal, Colorectal, Mesenteric, and Peritoneal Gastrointestinal Stromal Tumor AJCC v8
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Sarcoma | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Rogaratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (rogaratinib) (Experimental): Patients receive rogaratinib PO BID on days 1-28 of each cycle. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo biopsy at baseline and progression and CT, MRI, and PET-CT throughout the study. Patients may also undergo blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Rogaratinib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan and PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Rogaratinib — Given PO
  Other Names: BAY-1163877; BAY1163877

SUMMARY:
This phase II trial studies the effect of rogaratinib in treating patients with sarcoma with a change in a group of proteins called fibroblast growth factor receptors (FGFRs) or SDH-deficient gastrointestinal stromal tumor (GIST). Rogaratinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the objective radiographic response rate to single agent rogaratinib (BAY 1163877) in two cohorts of patients with sarcoma: Cohort A defined as patients with a sarcoma which harbors an alteration in fibroblast growth factor receptor (FGFR) 1, 2, 3 or 4 identified by next-generation sequencing profiling, and Cohort B defined as patients with advanced succinate dehydrogenase (SDH)-deficient gastrointestinal stromal tumor (GIST).

SECONDARY OBJECTIVES:

I. To estimate progression-free survival (PFS) in patients in Cohort A and Cohort B treated with rogaratinib (BAY 1163877).

II. Further assessment for safety and tolerability.

EXPLORATORY OBJECTIVES:

I. To evaluate serial measurements of FGFR and FGFR ligand in serial tumor biopsies as potential pharmacodynamic markers of FGFR pathway inhibition by ribonucleic acid sequencing (RNA-seq) (pre-treatment biopsy and post-progression biopsy [if available]).

II. Whole exome sequencing (WES) of the pre-treatment biopsy and post-progression biopsy (if available) to help identify mechanisms of resistance.

III. To bank tumor material, germline deoxyribonucleic acid (DNA), and peripheral blood for potential future research for participating subjects who provide additional consent.

IV. To explore rogaratinib exposure with pharmacodynamics effects (i.e., clinical response, toxicity, and markers of FGFR pathway inhibition).

OUTLINE:

Patients receive rogaratinib orally (PO) twice daily (BID) on days 1-28 of each cycle. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo biopsy at baseline and progression and computed tomography (CT), magnetic resonance imaging (MRI), and positron emission tomography (PET)-CT throughout the study. Patients may also undergo blood sample collection on study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically confirmed sarcoma with FGFR alteration identified by next-generation sequencing profiling with the exception of SDH-deficient GIST who can be enrolled regardless of FGFR status. Initial testing can be performed on archival tissue, if available. Patients must have locally advanced or metastatic disease that is not amenable to surgery
* Presence of measurable disease: Patient must have measurable disease
* Patients must have progressed following at least one standard prior chemotherapy regimen with the exception of SDH-deficient GIST for which there is no standard of care
* Participant must be willing to undergo pre-treatment biopsy if disease site is amenable to biopsy and low risk for the biopsy procedure. If biopsy is not possible, eligibility may be approved after discussion with the Study Chair. Of note, a minimum of 15 participants in each arm open to stage 2 should have disease amenable to biopsy. For those arms open in stage 1, all patients should have biopsiable disease.
* Age >= 18 years

  * Because no dosing or adverse event data are currently available on the use of rogaratinib (BAY 1163877) in patients <18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Hemoglobin >= 8.0 g/dL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3.0 x institutional ULN (unless liver metastases are present in which case it must be =< 5 x ULN)
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 (using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)
* Human immunodeficiency virus (HIV)-infected patients on effective non-CYP3A4 interacting anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients must be disease-free of prior invasive malignancies for > 5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix

  * NOTE: If there is a history of prior malignancy, patients must not be receiving other specific treatment for that cancer
* Patients should have completed prior treatment for their cancer: chemotherapy or radiotherapy must have been completed for greater than 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients should have recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class 2B or better
* Patients must have a QTc interval length of below 450 millisecond (msec)
* Participant is willing to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Participant must be able to swallow and maintain pills
* Women of childbearing potential must have a negative urine or serum pregnancy test within 28 days of initial dose of rogaratinib (BAY 1163877), and again within 7 days prior to treatment on day 1. If screening occurs within 7 days of day 1, only one pregnancy test is required
* The effects of rogaratinib (BAY 1163877) on the developing human fetus are unknown. For this reason and because kinase inhibitor agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of rogaratinib (BAY 1163877). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of rogaratinib (BAY 1163877) administration
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to rogaratinib (BAY 1163877)
* Concomitant administration with sensitive substrates/narrow therapeutic index drugs of CYP3A4, P-gp BCRP, MATE1, and MATE2K, and strong inhibitors and inducers of CYP3A4 should be avoided. Use caution with strong inhibitors and inducers of P-glycoprotein (gp). Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Concomitant administration of medications that prolong QT/QTc interval is prohibited in accordance with the published FDA guidance "E14 Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs".
* Patients with disturbed calcium and/or phosphate metabolism are excluded from this study
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because rogaratinib (BAY 1163877) is kinase inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with rogaratinib (BAY 1163877), breastfeeding should be discontinued if the mother is treated with rogaratinib (BAY 1163877)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective radiographic response | Up to 30 days after removal from study
  The duration of overall response is measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

SECONDARY OUTCOMES:
Progression-free survival | From start of treatment to time of progression or death, whichever occurs first, assessed up to 30 days after removal from study
  Will be estimated using Kaplan-Meier method.
Incidence of adverse events | Up to 30 days after removal from study
  Adverse events will be measured by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

OTHER OUTCOMES:
Serial measurements of FGFR and FGFR ligand | Up to 30 days after removal from study
  Will be evaluated in serial tumor biopsies as potential pharmacodynamic markers of FGFR pathway inhibition by ribonucleic acid sequencing. Estimation of continuous biomarker measures will be via mean or median as appropriate and standard deviation.
Mechanisms of resistance | Up to 30 days after removal from study
  Will identify mechanisms of resistance via whole exome sequencing of pre- and post-treatment biopsies and considered exploratory.
Banking of tumor material, germline deoxyribonucleic acid, and peripheral blood | Up to 30 days after removal from study
  Will be banked for potential research.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne George, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (18):
- United States (18):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Northwestern University, Chicago, Illinois
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/47/NCT04595747/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/47/NCT04595747/ICF_001.pdf